CLINICAL TRIAL: NCT05702606
Title: Radial Extracorporeal Shock Wave Therapy for Management of Spasticity in Patients With Cerebral Palsy
Brief Title: Shock Wave Therapy for Management of Spasticity in Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Aspace Catalunya (Other)
Responsible Party: Principal Investigator, Míriam Tur, Principal Investigator, Fundacio Aspace Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASP_Shock_MT
Record Dates: First submitted 2022-11-29; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy; Spasticity, Muscle; Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): 3 rESWT sessions with a time interval of 1 week between each session.
  Interventions: Other: Radial extracorporeal shock wave therapy (rESWT)
- Experimental Group A (Experimental): 3 rESTW sessions with a time interval of 2 weeks between each session.
  Interventions: Other: Radial extracorporeal shock wave therapy (rESWT)
- Experimental Group B (Experimental): 3 rESTW sessions with a time interval of 4 weeks between each session.
  Interventions: Other: Radial extracorporeal shock wave therapy (rESWT)

INTERVENTIONS:
Other: Radial extracorporeal shock wave therapy (rESWT) — Radial shock waves are ballistic waves generated by injection of compressed air inside an applicator that fires a projectile into the itself and impacts against the application head

SUMMARY:
Spasticity is the most common motor disorder in cerebral palsy (CP). The objectives of his therapeutic approach include; reducing pain, ease of use of orthopedic aids, improving posture, minimizing contractures and deformity, and facilitating mobility and dexterity, with the ultimate goal of maximizing the potential of the patient and promoting their independence and quality of life. The approach to spasticity in CP is complex and presents itself as a great challenge for the rehabilitation team. Radial extracorporeal shock wave therapy (rESWT) has been established in recent years as an effective, non-invasive alternative with hardly any side effects (small bruises or discomfort during the application) for the management of spasticity in patients with CP. rESWT is a relatively new therapy in the field of neurology, in 2010 was published the first clinical trial where shock waves were applied for the management of spasticity in patients with CP. Currently, few works have studied the efficacy of rESWT in patients with CP. In all of them, the results demonstrated the treatment's effectiveness in reducing spasticity locally in people with CP up to 3 months after the application. The group most studied muscle has been the Triceps Surae, and there is a great disparity regarding the doses of treatment applied in each study, especially regarding the number of sessions and the time interval between sessions. The most widely used protocol is 3 rESWT sessions with a time interval of 1 week between session; This protocol was established as the most effective in the treatment of trauma pathology. Despite all the variability in the administration of the dose, we have been able to observe that none of them has studied the effect of rESWT by lengthening the time interval between sessions beyond one week to check whether the therapeutic effects on spasticity can be prolonged over time by applying the same dose. Most of the studies conclude that future research should be aimed at studying the most optimal dose of treatment as well as evaluating the long-term results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP.
* With a CP classified as spastic.
* Spasticity in the Triceps Surae muscle.
* Who have a Gross Motor Classification (GMFCS) level between l and ll
* Having signed the informed consent by the participant or your legal guardian

Exclusion Criteria:

* Have received treatment with shock waves in the Triceps Surae or any other muscle of the lower extremity in the 6 months before the study.
* Have received treatment with botulinum toxin and/or treatment focal intramuscular injection with phenol or alcohol in the Triceps Surae or some other lower extremity muscle in the 6 months before the study.
* Patients who have undergone surgery for deformities foot orthotics in the last year.
* Fixed deformities in the ankle joint.
* Clinical signs of myopathy and neuropathy.
* Infection or tumor at the site of application of the therapy*.
* Severe blood dyscrasia*.
* Blood coagulation disorders*.
* Treatment with oral anticoagulants*

  * Contraindications of radial extracorporeal shock wave therapy.

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Change in passive range of movement and the stretching reflex in ankle dorsiflexion. Tardieu Scale | Base line,3,5,9,12 and 24 weeks
  Assess the change in degrees of passive range of motion and the ankle dorsiflexion stretch reflex measured with an inclinometer
Change in goal attainment scale (GAS) | Setting of goal(s) at start (base line), assesment al 3,5,9,12 and 24 weeks
  Goal attainment scale: Definition of an individual goal at the start. Will be assess the achievement or not of an objective and evaluates the expectations of improvement in each of the goals with a numerical scale from -2 to +2:
  (-2) Result much lower than expected (-1) Lower than expected result (0) Expected result (+1) Result higher than expected (+2) Result much higher than expected

SECONDARY OUTCOMES:
Pain secondary to spasticity assessed by the visual analog scale | Base line,3,5,9,12 and 24 weeks
  If the patient presents pain secondary to spasticity, evaluate the degree of improvement after therapy using the visual analog scale where the value 0 is no pain and 10 is the worst possible pain.
Satisfaction with the therapy assessed by the visual analog scale | Base line,3,5,9,12 and 24 weeks
  Evaluate the degree of improvement perceived by the patient in relation to the therapy using the visual analog scale where the value 0 is no perceived improvement and 10 is the maximum expected improvement
Adverse effects by Data collection notebook | Base line,3,5,9,12 and 24 weeks
  Possible adverse effects secondary to treatment such as small bruises, petechiae, or muscle fatigue will be recorded in the data collection notebook

CONTACTS AND LOCATIONS:
Overall Officials: Míriam Tur Segura, First, Principal Investigator — Fundació Aspace Catalunya; Raimon Milà Villarroel, third, Study Director — Facultat de Ciències de la Salut Blanquerna - Universitat Ramon Llull
Locations (1):
- Fundació Aspace Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society; Delgado MR, Hirtz D, Aisen M, Ashwal S, Fehlings DL, McLaughlin J, Morrison LA, Shrader MW, Tilton A, Vargus-Adams J. Practice parameter: pharmacologic treatment of spasticity in children and adolescents with cerebral palsy (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2010 Jan 26;74(4):336-43. doi: 10.1212/WNL.0b013e3181cbcd2f. PMID 20101040
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Spasticity in Children and Young People with Non-Progressive Brain Disorders: Management of Spasticity and Co-Existing Motor Disorders and Their Early Musculoskeletal Complications. London: RCOG Press; 2012 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK116583/ PMID 23346608
- [Background] Ramstad K, Jahnsen R, Skjeldal OH, Diseth TH. Characteristics of recurrent musculoskeletal pain in children with cerebral palsy aged 8 to 18 years. Dev Med Child Neurol. 2011 Nov;53(11):1013-8. doi: 10.1111/j.1469-8749.2011.04070.x. PMID 22014321
- [Background] Benini R, Shevell MI. Updates in the treatment of spasticity associated with cerebral palsy. Curr Treat Options Neurol. 2012 Dec;14(6):650-9. doi: 10.1007/s11940-012-0192-7. PMID 22851256
- [Background] Ogden JA, Alvarez RG, Levitt R, Marlow M. Shock wave therapy (Orthotripsy) in musculoskeletal disorders. Clin Orthop Relat Res. 2001 Jun;(387):22-40. doi: 10.1097/00003086-200106000-00005. PMID 11400888
- [Background] Schmitz C, Csaszar NB, Milz S, Schieker M, Maffulli N, Rompe JD, Furia JP. Efficacy and safety of extracorporeal shock wave therapy for orthopedic conditions: a systematic review on studies listed in the PEDro database. Br Med Bull. 2015;116(1):115-38. doi: 10.1093/bmb/ldv047. Epub 2015 Nov 18. PMID 26585999
- [Background] Mattyasovszky SG, Langendorf EK, Ritz U, Schmitz C, Schmidtmann I, Nowak TE, Wagner D, Hofmann A, Rommens PM, Drees P. Exposure to radial extracorporeal shock waves modulates viability and gene expression of human skeletal muscle cells: a controlled in vitro study. J Orthop Surg Res. 2018 Apr 6;13(1):75. doi: 10.1186/s13018-018-0779-0. PMID 29625618
- [Background] Manganotti P, Amelio E. Long-term effect of shock wave therapy on upper limb hypertonia in patients affected by stroke. Stroke. 2005 Sep;36(9):1967-71. doi: 10.1161/01.STR.0000177880.06663.5c. Epub 2005 Aug 18. PMID 16109905
- [Background] Amelio E, Manganotti P. Effect of shock wave stimulation on hypertonic plantar flexor muscles in patients with cerebral palsy: a placebo-controlled study. J Rehabil Med. 2010 Apr;42(4):339-43. doi: 10.2340/16501977-0522. PMID 20358168
- [Background] Vidal X, Morral A, Costa L, Tur M. Radial extracorporeal shock wave therapy (rESWT) in the treatment of spasticity in cerebral palsy: a randomized, placebo-controlled clinical trial. NeuroRehabilitation. 2011;29(4):413-9. doi: 10.3233/NRE-2011-0720. PMID 22207070
- [Background] Vidal X, Marti-Fabregas J, Canet O, Roque M, Morral A, Tur M, Schmitz C, Sitja-Rabert M. Efficacy of radial extracorporeal shock wave therapy compared with botulinum toxin type A injection in treatment of lower extremity spasticity in subjects with cerebral palsy: A randomized, controlled, cross-over study. J Rehabil Med. 2020 Jun 30;52(6):jrm00076. doi: 10.2340/16501977-2703. PMID 32556354
- [Derived] Tur Segura M, Gimeno Esteve F, Biedermann Villagra T, Jimenez Redondo J, Garcia Rodriguez N, Mila Villarroel R. Radial extracorporeal shock wave therapy for the management of spasticity in cerebral palsy: study protocol for a randomized controlled trial. Front Neurol. 2024 Jun 13;15:1402452. doi: 10.3389/fneur.2024.1402452. eCollection 2024. PMID 38957349